CLINICAL TRIAL: NCT03221634
Title: A Phase 2 Study of Pembrolizumab in Combination With Daratumumab (Anti CD38) in Participants With Relapsed Refractory Multiple Myeloma (rrMM)
Brief Title: Efficacy and Safety Study of Pembrolizumab (MK-3475) in Combination With Daratumumab in Participants With Relapsed Refractory Multiple Myeloma (MK-3475-668/KEYNOTE-668)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-668; 2017-001001-32 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Multiple Myeloma
Keywords: Programmed cell death 1 receptor (PD1); PD-1; Programmed cell death ligand 1 receptor (PDL1); PD-L1
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg by intravenous (IV) infusion once every 3 weeks (Q3W) for up to 35 administrations (up to approximately 2 years) and receive daratumumab 16 mg/kg by IV infusion on Days 1, 8, 15, and 22 of Cycles 1-2; on Days 1 and 15 of Cycles 3-6, and on Day 1 of Cycle 7 and beyond, for up to 2 years. Each cycle is 28 days long.
  Interventions: Biological: Pembrolizumab; Biological: Daratumumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475
Biological: Daratumumab — IV infusion
  Other Names: DARZALEX®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of pembrolizumab (MK-3475) in combination with daratumumab in participants with relapsed refractory multiple myeloma (rrMM). The primary outcome measure for this study is the assessment of Objective Response Rate (ORR) in participants with rrMM.

DETAILED DESCRIPTION:
Study treatment will continue until the participant has completed 35 infusions (approximately 2 years) of pembrolizumab treatment. All participants who stop study treatment with stable disease (SD) or better may be eligible for up to an additional ~1 year of study treatment if they progress after stopping study treatment from the initial treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of active MM and measurable disease defined as: a.) Serum M-protein levels ≥0.5 g/dL or b.) Urine M-protein levels ≥200 mg/24 hours or c.) For participants without measurable serum and urine M-protein levels, an abnormal serum free light chain ratio (FLC κ/λ) with involved FLC level ≥100 mg/L.
* Has undergone prior treatment with ≥2 treatment lines of anti-myeloma therapy and must have failed their last line of treatment defined as lack of response or documented disease progression during or within 60 days of completing their last anti-myeloma therapy.
* Prior anti-myeloma treatments must have included an immunomodulatory drug (IMiD; i.e., lenalidomide, thalidomide, or pomalidomide) AND a proteasome inhibitor (PI; i.e., bortezomib, ixazomib, or carfilzomib) alone or in combination and participant must have failed therapy with an IMiD or PI or both.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Has adequate organ function.
* Male participants must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants must not be pregnant, breastfeeding, and must agree to use (or have their partner use) acceptable contraception during heterosexual activity during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

* Has oligo-secretory myeloma, smoldering multiple myeloma (SMM), monoclonal gammopathy of undetermined significance (MGUS), Waldenström's macroglobulinemia, or any history of plasma cell leukemia.
* Has a history of repeated infections, primary amyloidosis, hyperviscosity, or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include early stage cancers (carcinoma in situ or Stage 1) treated with curative intent, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer, or in situ breast cancer that has undergone potentially curative therapy.
* Has known meningeal involvement of MM.
* Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or daratumumab and any of its excipients.
* Has known allergies, hypersensitivity, or intolerance to monoclonal antibodies (mAbs) or human proteins, or their excipients, or known sensitivity to mammalian-derived products.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has either of the following: a.) Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal, or b.) Known moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of hepatitis B or known active hepatitis C.
* Has a known history of active tuberculosis (TB).
* Has received prior solid organ transplant.
* Has clinically significant cardiac disease or electrocardiogram (ECG) abnormalities or any history of clinically significant ventricular arrhythmias.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
* Has previously received daratumumab or other anti-cluster of differentiation 38 (anti-CD38) therapies.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (i.e., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137) or has previously participated in a Merck pembrolizumab (MK-3475) clinical study.
* Has received prior anti-myeloma therapy including but not limited to dexamethasone, IMiDs, PIs, monoclonal antibody, chemotherapy, or radiation therapy within 4 weeks or 5 half-lives (whichever is longer) before first dose of study treatment or not recovered (≤ Grade 1 or at Baseline) from AEs due to previously administered agents.
* Has undergone prior allogeneic stem cell transplant (allo-SCT) within the last 5 years.
* Has received autologous stem cell transplant (auto-SCT) within 12 weeks before the first dose of study treatment or are planning for or are eligible for auto- or allo-SCT.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-03-20 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants who experience a partial response (PR; ≥50% reduction of serum myeloma (M)-protein plus reduction in 24-hour urinary M-protein by ≥90% or to <200 mg per 24 hours) or better per International Myeloma Working Group (IMWG) 2016, based on investigator assessment.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants who experience stable disease (SD; not meeting criteria for complete response, very good partial response, partial response, minimal response or progressive disease) or better prior to any evidence of progression, per IMWG 2016 based on investigator assessment.
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from first documented evidence of at least a PR (≥50% reduction of serum M-protein plus reduction in 24-hour urinary M-protein by ≥90% or to <200 mg per 24 hours) until disease progression or death, per IMWG 2016, based on investigator assessment.
Adverse Events (AEs) | Up to approximately 27 months
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing one or more AEs will be assessed.
Study Treatment Discontinuations Due to AEs | Up to approximately 2 years
  The number of participants discontinuing study treatment due to AEs will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (23):
- United States (3):
  - Mayo Clinic Jacksonville ( Site 0003), Jacksonville, Florida
  - Emory University School of Medicine ( Site 0002), Atlanta, Georgia
  - Karmanos Cancer Institute ( Site 0001), Bloomfield Hills, Michigan
- Canada (6):
  - Calgary Lab Services - Foothills Medical Centre ( Site 0105), Calgary, Alberta
  - Cross Cancer Institute ( Site 0104), Edmonton, Alberta
  - Capital Health Queen Elizabeth II Health Sciences Centre ( Site 0101), Halifax, Nova Scotia
  - Hopital Maisonneuve-Rosemont [Montreal, Canada] ( Site 0102), Montreal, Quebec
  - McGill University Health Centre ( Site 0100), Montreal, Quebec
  - CHU de Quebec - Hopital de l'Enfant-Jesus ( Site 0106), Québec, Quebec
- France (3):
  - CHRU Lille Hospital Claude Huriez ( Site 0200), Lille
  - Hopital Saint-Louis ( Site 0202), Paris
  - Centre Hopitalier Lyon Sud ( Site 0201), Pierre-Bénite
- Israel (4):
  - Rambam Medical Center ( Site 0700), Haifa
  - Rabin Medical Center ( Site 0702), Petah Tikva
  - Sourasky Medical Center ( Site 0701), Tel Aviv
  - Sheba MC ( Site 0703), Tel Litwinsky
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol ( Site 0302), Badalona
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 0303), L'Hospitalet de Llobregat
  - Clinica Universitaria de Navarra ( Site 0301), Pamplona
  - Hospital Clinico Universitario de Salamanca ( Site 0300), Salamanca
  - Hospital Clinico Universitario de Valencia ( Site 0304), Valencia
- Sweden (2):
  - Skaenes Universitetssjukhus Lund ( Site 0500), Lund
  - Karolinska Universitetssjukhuset ( Site 0501), Stockholm